CLINICAL TRIAL: NCT01605487
Title: Double-blind, Three-way Cross-over, Placebo-controlled Study to Assess the Efficacy, Safety and Mechanisms of Treatment With Rupatadine 20 mg and 40 mg in Cold Contact Urticaria (CCU)
Brief Title: Study to Assess Efficacy, Safety and Mechanism of Rupatadine in Cold Urticaria
Acronym: PAFCUTIII
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Charite University, Berlin, Germany (Other)
Collaborators: Hospital del Mar (Other)
Responsible Party: Principal Investigator, Marina Abajian, MD, Charite University, Berlin, Germany
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: PAFCUTIII
Record Dates: First submitted 2012-05-11; First posted 2012-05-25 (Estimated); Last update posted 2014-10-15 (Estimated); Status verified 2014-04

CONDITIONS: Cold Contact Urticaria
MeSH Terms: conditions — Cold Urticaria | interventions — rupatadine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (6):
- Rupatadine 20mg - Placebo - Rupatadine 40mg (Other)
  Interventions: Drug: Rupatadine
- Rupatadine 20mg - Rupatadine 40mg - Placebo (Other)
  Interventions: Drug: Rupatadine
- Placebo - Rupatadine 20mg - Rupatadine 40mg (Other)
  Interventions: Drug: Rupatadine
- Rupatadine 40mg - Placebo - Rupatadine 20mg (Other)
  Interventions: Drug: Rupatadine
- Placebo - Rupatadine 40mg - Rupatadine 20mg (Other)
  Interventions: Drug: Rupatadine
- Rupatadine 40mg - Rupatadine 20mg - Placebo (Other)
  Interventions: Drug: Rupatadine

INTERVENTIONS:
Drug: Rupatadine — Rupatadine in Tab 10mg: 4 Tab.(2 Tab. of Rupatadine + 2 Tab. of Placebo) once daily during 7 days, then 14 days washout period; Placebo 4 Tab once daily during 7 days, then 14 days washout period; Rupatadine in Tab. 10mg, 4 Tab. once daily during 7 days
  Arms: Rupatadine 20mg - Placebo - Rupatadine 40mg
Drug: Rupatadine — Rupatadine in Tab 10mg: 4 Tab.(2 Tab. of Rupatadine + 2 Tab. of Placebo) once daily during 7 days, then 14 days washout period; Rupatadine in Tab. 10mg, 4 Tab. once daily during 7 days,then 14 days washout period; Placebo 4 Tab once daily during 7 days
  Arms: Rupatadine 20mg - Rupatadine 40mg - Placebo
Drug: Rupatadine — Placebo 4 Tab once daily during 7 days, then 14 days washout period; Rupatadine in Tab 10mg: 4 Tab.(2 Tab. of Rupatadine + 2 Tab. of Placebo) once daily during 7 days, then 14 days washout period; Rupatadine in Tab. 10mg, 4 Tab. once daily during 7 days
  Arms: Placebo - Rupatadine 20mg - Rupatadine 40mg
Drug: Rupatadine — Rupatadine in Tab. 10mg, 4 Tab. once daily during 7 days,then 14 days washout period; Placebo 4 Tab once daily during 7 days, then 14 days washout period; Rupatadine in Tab 10mg: 4 Tab.(2 Tab. of Rupatadine + 2 Tab. of Placebo) once daily during 7 days
  Arms: Rupatadine 40mg - Placebo - Rupatadine 20mg
Drug: Rupatadine — Placebo 4 Tab once daily during 7 days, then 14 days washout period; Rupatadine in Tab. 10mg, 4 Tab. once daily during 7 days, then 14 days washout period; Rupatadine in Tab 10mg: 4 Tab.(2 Tab. of Rupatadine + 2 Tab. of Placebo) once daily during 7 days
  Arms: Placebo - Rupatadine 40mg - Rupatadine 20mg
Drug: Rupatadine — Rupatadine in Tab. 10mg: 4 Tab. once daily during 7 days, then 14 days washout period; Rupatadine in Tab 10mg: 4 Tab.(2 Tab. of Rupatadine + 2 Tab. of Placebo) once daily during 7 days, then 14 days washout period; Placebo 4 Tab once daily during 7 days
  Arms: Rupatadine 40mg - Rupatadine 20mg - Placebo

SUMMARY:
Main objective of this study is to evaluate the efficacy of rupatadine in 20 mg and 40 mg doses in the development of symptoms of cold contact urticaria. For this purpose, a Peltier element-based electronic provocation device (TempTest®, emo systems GmbH, Berlin, Germany) will be used. This allows skin exposure to 12 different temperatures from 4 to 42 °C simultaneously in a standardized and reproducible way and thus the determination of individual temperature and/or stimulation time thresholds.

In addition mediators related from activated must cells such as histamine, PAF, PGD2 should be identified in the period between the application of stimulus and the appearance of symptoms of cold urticaria and should be characterized qualitatively and quantitatively.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent signed and dated
* Reliable method of contraception for both women of childbearing potential as well as man during the study and 3 months thereafter. A highly effective method of birth control is defined as those which result in a low failure rate (i.e. less than 1% per year) when used consistently and correctly such as implants, injectables, combined oral contraceptives, some IUDs, sexual abstinence or vasectomised partner
* Outpatients with CCU for more than 6 weeks. Urticaria symptoms must comprise wheal and itch after contact cooling of the skin. Provocation should be performed by application of Temptest®3.0 which allows for reproducible and standardized cold provocation tests and the identification of temperature and stimulation time thresholds.
* Age 18 and above 18 years.
* No participation in other clinical trials 1 months before and after participation in this study

Exclusion Criteria:

* Subjects who are inmates of psychiatric wards, prisons, or other state institutions. Existing or planned placement in an institution after ruling according to § 40 passage 1, number 4 AMG (Arzneimittelgesetz).
* The presence of permanent severe diseases, especially those affecting the immune system, except urticaria and cold urticaria
* The presence of permanent gastrointestinal condition which may influence the oral therapy (chronic diarrhoea diseases, congenital malformations or surgical mutilations of gastrointestinal tract)
* History or presence of epilepsy, significant neurological disorders, cerebrovascular attacks or ischemia
* History or presence of myocardial infarction or cardiac arrhythmia which requires drug therapy
* ECG alterations of repolarisation (QTc prolongations > 450ms)
* Blood pressure >180/100 mmHg and/or heart rate >100/min.
* Evidence of significant hepatic or renal disease (GOT and/or GPT 3 times above the upper reference value, serum creatinine 1.5 times above the upper reference value)
* History of hypersensitivity or allergic reaction to rupatadine or its ingredients or any other antihistamine compounds.
* Presence of active cancer which requires chemotherapy or radiation therapy
* Presence of lactose and galactose intolerance or with glucose-galactose malabsorption
* Simultaneous chronic spontaneous or physical urticaria that could interfere CCU clinical assessment
* Intake of antihistamines or antileukotrienes within 7 days before beginning of the study
* Intake of oral or depot corticosteroids within 14 days prior to screening visit
* Use of systemic immunosupressants/immunomodulators like cyclosporine A, dapsone, methotrexate, mycophenolate, chloroquine, and comparable drugs within 28 days prior to screening visit.
* Use of ketoconazole, erythromycin or potential inhibitors of the isoenzyme CYP3A4 of the cytochrome P450.
* Currently abusing drugs or alcohol
* Unwilling or unable to comply with the protocol
* Pregnancy or breast-feeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2012-06; Primary Completion 2013-09 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Critical stimulation time threshold(CSTT) after challenge with cold | Visit 1(day -14 Screening), Visit 2 (Randomization; day 0), Visit 3(Last day of treatment period 1; day 7), Visit 4(Last day of treatment period 2; day 28), Visit 5(Last day of treatment period 3; day 49)
  Critical stimulation time threshold (CSTT) determines the shortest stimulation time sufficient for inducing a wheal-and-flare reaction
Critical temperature threshold (CTT)after challenge with cold | Visit 1(day -14 Screening), Visit 2 (Randomization; day 0), Visit 3(Last day of treatment period 1; day 7), Visit 4(Last day of treatment period 2; day 28), Visit 5(Last day of treatment period 3; day 49)
  Critical temperature threshold (CTT) determines the highest temperature sufficient for inducing a wheal-and-flare reaction

SECONDARY OUTCOMES:
Mast cell mediator release | Visit 3(Last day of treatment period 1; day 7), Visit 4(Last day of treatment period 2; day 28), Visit 5(Last day of treatment period 3; day 49)
Safety and tolerability following administration of Rupatadine to patients with cold contact urticaria | up to 9 weeks
  Safety and tolerability: This includes physical examination, routine safety laboratory assessments, clinical observation, vital sings and adverse event reporting

CONTACTS AND LOCATIONS:
Overall Officials: Karoline Krause, MD, Principal Investigator — Charite University, Berlin, Germany
Locations (1):
- Department of Dermatology and Allergy, Charité - Universitätsmedizin Berlin, Charitéplatz 1, Germany